CLINICAL TRIAL: NCT00049842
Title: PEG-Intron(TM) Maintenance Therapy vs. an Untreated Control Group for Prevention of Progression of Fibrosis in Adult Subjects With Chronic Hepatitis C With Hepatic Fibrosis (METAVIR Fibrosis Score of F2 or F3), Who Failed Therapy With PEG-Intron Plus REBETOL(R) (in Protocol No. P02370)
Brief Title: Prevention of Disease Progress in Chronic Hepatitis C Patients With Liver Fibrosis (Study P02570AM2)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P02570
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Chronic Hepatitis C; Liver Fibrosis
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG-Intron (peginterferon alfa-2b) 0.5 µg/kg Weekly (QW) (Experimental): PEG-Intron 0.5 µg/kg Weekly (QW) subcutaneously (SC) as maintenance therapy for 36 months with 4-week follow-up
  Interventions: Biological: peginterferon alfa-2b (SCH 54031)
- Untreated Control (No Intervention)

INTERVENTIONS:
Biological: peginterferon alfa-2b (SCH 54031) — 0.5 µg/kg Weekly QW SC for 36 months
  Arms: PEG-Intron (peginterferon alfa-2b) 0.5 µg/kg Weekly (QW)

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of PEG-Intron versus no treatment for the prevention of fibrosis progression in adult participants with moderate to severe liver fibrosis secondary to chronic hepatitis C, who failed PEG-Intron plus Rebetol treatment in protocol P02370 (NCT00039871).

ELIGIBILITY:
Inclusion Criteria:

* Age at entry in study P02370 (NCT00039871) 18-65 years;
* Nonresponder to PEG-Intron plus Rebetol in study P02370

Exclusion Criteria:

* Participants who did not participate in the P02370 study.
* Any medical condition, including but not limited to decompensated liver disease, malignancy or substance abuse, that developed during the P02370 study which could interfere with the participant's participation in and completion of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2002-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Poynard T, Bruix J, Schiff ER, Diago M, Berg T, Moreno-Otero R, Lyra AC, Carrilho F, Griffel LH, Boparai N, Jiang R, Burroughs M, Brass CA, Albrecht JK. Improved inflammatory activity with peginterferon alfa-2b maintenance therapy in non-cirrhotic prior non-responders: a randomized study. J Hepatol. 2013 Mar;58(3):452-9. doi: 10.1016/j.jhep.2012.11.001. Epub 2012 Nov 14. PMID 23159770

RESULTS

PARTICIPANT FLOW:
Groups:
- Untreated Control: Participants were observed (no treatment given) for 36 months with 4-week follow-up
Period: Treatment Phase
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control
Started | 270 | 270
Completed | 177 | 192
Not Completed | 93 | 78
Not completed — Adverse Event | 47 | 12
Not completed — Withdrawal by Subject | 35 | 46
Not completed — Non-compliance with protocol | 7 | 8
Not completed — Lost to Follow-up | 4 | 8
Not completed — Administrative | 0 | 3
Not completed — Did not meet protocol eligibility | 0 | 1
Period: Follow-up Phase
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control
Started | 218 (Population is all treatment phase completers plus some who discontinued the treatment phase.) | 194 (Population is all treatment phase completers plus some who discontinued the treatment phase.)
Completed | 211 | 189
Not Completed | 7 | 5
Not completed — Adverse Event | 6 | 1
Not completed — Other | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control | Total
Number analyzed (Participants) | 270 | 270 | 540
Age, Customized [Number; unit: participants]
  <=50 years | 145 | 148 | 293
  >50 years | 125 | 122 | 247
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 81 | 157
  Male | 194 | 189 | 383

OUTCOME MEASURES:

1. Primary Outcome: Fibrosis Response Status (ie, Improvement, no Change, or the Worsening of the Fibrosis Score in Participants With Baseline METAVIR Fibrosis Score of F2 or F3).
Description: Definitions:
  Fibrosis scoring: F0 (no fibrosis), F1 (stellate enlargement of portal tract without septa formation, F2 (enlargement of portal tract with rare septa formation, F3 (numerous septa without cirrhosis), F4 (cirrhosis).
  Improved: Participants whose METAVIR fibrosis score at up to Month-36 decreases by 1 or more units compared to baseline.
  No Change: Participants whose METAVIR fibrosis score at up to Month-36 is the same as the baseline score.
  Worsened: Participants whose METAVIR fibrosis score at up to Month-36 increases by 1 or more units compared to baseline.
Time Frame: Baseline to up to Month-36
Population: Population is Intent-to-Treat (ITT). Participants with missing Month-36 biopsy slides were classified as "no change", including 88 participants in the PEG-Intron group and 104 participants in the Observed group.
Measure: Number; unit: Participants
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control
Number analyzed (Participants) | 270 | 270
Participants
  Improved | 44 | 29
  No Change | 162 | 176
  Worsened | 64 | 65

2. Secondary Outcome: Inflammation Response Status (ie, Improvement, no Change, or the Worsening of the METAVIR Activity Score as Compared to Baseline)
Description: Activity Scoring: A0 (no histological activity), A1 (minimal activity), A2 (moderate activity), A3 (severe activity), A4 (lobular chronic hepatitis).
  Changes in liver inflammation defined as follows:
  Improved: Participants whose METAVIR activity score at up to Month-36 decreases by 1 or more units compared to baseline.
  No Change: Participants whose METAVIR activity score at up to Month-36 is the same as the baseline score.
  Worsened: Participants whose METAVIR activity score at up to Month-36 increases by 1 or more units compared to baseline.
Time Frame: Baseline to up to Month-36
Population: Population is ITT. Participants with missing Month-36 biopsy slides were classified as "no change", including 88 participants in the PEG-Intron group and 104 participants in the Observed group.
Measure: Number; unit: Participants
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control
Number analyzed (Participants) | 270 | 270
Participants
  Improved | 54 | 23
  No Change | 195 | 209
  Worsened | 21 | 38

3. Secondary Outcome: Mean Change From Baseline to up to Month-36 in the METAVIR Fibrosis Score (Using a Continuous Scale)
Description: The change of Metavir Fibrosis Score = Metavir Fibrosis Score at up to Month-36 - Metavir Fibrosis Score at Baseline.
  Fibrosis scoring: 0 (no fibrosis), 1 (stellate enlargement of portal tract without septa formation, 2 (enlargement of portal tract with rare septa formation, 3 (numerous septa without cirrhosis), 4 (cirrhosis).
Time Frame: Baseline to up to Month-36
Population: ITT population who had both pre and up to Month-36 METAVIR fibrosis score.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control
Number analyzed (Participants) | 182 | 166
Units on a scale | 0.13 (0.977) | 0.31 (1.002)

4. Secondary Outcome: The Number of Participants Whose METAVIR Fibrosis Score Did Not Worsen (ie, the Response Status of Improved/no Change) During Treatment Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline to up to Month-36
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control
Number analyzed (Participants) | 270 | 270
Participants
  Improved/No Change | 206 | 205
  Worsened | 64 | 65

5. Secondary Outcome: Mean Change in the METAVIR Activity Score (Using a Continuous Scale)
Description: The change of Metavir Activity Score = Metavir Activity Score at up to Month-36 - Metavir Activity Score at Baseline.
  Activity Scoring: 0 (no histological activity), 1 (minimal activity), 2 (moderate activity), 3 (severe activity), 4 (lobular chronic hepatitis).
Time Frame: Baseline to up to Month-36
Population: ITT population who had both pre and up to Month-36 METAVIR activity score.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control
Number analyzed (Participants) | 182 | 166
Units on a scale | -0.20 (0.709) | 0.11 (0.642)

6. Secondary Outcome: Number of Participants With no Worsening (ie, the Response Status of Improved/ no Change) in the METAVIR Activity Score During the Treatment.
Description: Definitions:
  Activity Scoring: A0 (no histological activity), A1 (minimal activity), A2 (moderate activity), A3 (severe activity), A4 (lobular chronic hepatitis).
  Improved: Participants whose METAVIR activity score at up to Month-36 decreases by 1 or more units compared to baseline.
  No Change: Participants whose METAVIR activity score at up to Month-36 is the same as the baseline score.
  Worsened: Participants whose METAVIR activity score at up to Month-36 increases by 1 or more units compared to baseline.
Time Frame: Baseline to up to Month-36
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PEG-Intron (Peginterferon Alfa-2b) 0.5 µg/kg Weekly (QW) | Untreated Control
Number analyzed (Participants) | 270 | 270
Participants
  Improved/No Change | 249 | 232
  Worsened | 21 | 38

ADVERSE EVENTS:
Arm/Group | PEG-Intron | Untreated Control
Serious Adverse Events (participants affected / at risk) | 53/270 | 31/270
Other Adverse Events (participants affected / at risk) | 234/270 | 200/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron (N=270) | Untreated Control (N=270)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC AMYLOIDOSIS (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY OSTIAL STENOSIS (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 0 (0) | 2 (2)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 (3) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0)
RETROPERITONEAL FIBROSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 1 (1)
CHEST PAIN (General disorders) | 3 (3) | 1 (1)
DISEASE PROGRESSION (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1)
HERNIA (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 2 (2)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 2 (2) | 0 (0)
CRYOGLOBULINAEMIA (Immune system disorders) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 2 (2) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 (2) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 2 (2) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
NARCOTIC INTOXICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SKIN INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PATELLOFEMORAL PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PLICA SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BURKITT'S LYMPHOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
COMA (Nervous system disorders) | 1 (1) | 0 (0)
HEMIPLEGIA (Nervous system disorders) | 1 (1) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1)
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (2) | 3 (3)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 2 (2)
GLOMERULONEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 (0) | 1 (3)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 2 (2)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURIGO (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SUBSTANCE ABUSER (Social circumstances) | 1 (1) | 0 (0)
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0)
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
ILIAC ARTERY STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (1)
VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-Intron (N=270) | Untreated Control (N=270)
NEUTROPENIA (Blood and lymphatic system disorders) | 32 (98) | 15 (20)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 18 (39) | 5 (10)
HYPOTHYROIDISM (Endocrine disorders) | 20 (25) | 5 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 (18) | 14 (17)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 22 (23) | 22 (30)
DIARRHOEA (Gastrointestinal disorders) | 28 (40) | 16 (22)
DYSPEPSIA (Gastrointestinal disorders) | 18 (19) | 22 (26)
NAUSEA (Gastrointestinal disorders) | 23 (28) | 16 (16)
ASTHENIA (General disorders) | 46 (92) | 30 (38)
CHILLS (General disorders) | 14 (17) | 3 (3)
FATIGUE (General disorders) | 66 (82) | 59 (68)
INFLUENZA LIKE ILLNESS (General disorders) | 34 (59) | 4 (4)
INJECTION SITE ERYTHEMA (General disorders) | 18 (219) | 0 (0)
INJECTION SITE REACTION (General disorders) | 17 (17) | 1 (1)
IRRITABILITY (General disorders) | 32 (43) | 13 (13)
PYREXIA (General disorders) | 30 (94) | 12 (13)
HEPATOMEGALY (Hepatobiliary disorders) | 9 (11) | 16 (17)
NASOPHARYNGITIS (Infections and infestations) | 19 (26) | 14 (24)
DECREASED APPETITE (Metabolism and nutrition disorders) | 21 (26) | 10 (11)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 50 (79) | 40 (47)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 32 (46) | 24 (41)
MYALGIA (Musculoskeletal and connective tissue disorders) | 46 (228) | 20 (22)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 16 (18) | 9 (10)
DIZZINESS (Nervous system disorders) | 15 (21) | 11 (11)
HEADACHE (Nervous system disorders) | 76 (429) | 24 (31)
ANXIETY (Psychiatric disorders) | 25 (34) | 25 (35)
DEPRESSION (Psychiatric disorders) | 33 (41) | 24 (34)
INSOMNIA (Psychiatric disorders) | 56 (88) | 46 (58)
COUGH (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 16 (19)
ALOPECIA (Skin and subcutaneous tissue disorders) | 38 (43) | 21 (21)
DRY SKIN (Skin and subcutaneous tissue disorders) | 26 (29) | 7 (7)
PRURITUS (Skin and subcutaneous tissue disorders) | 36 (42) | 16 (17)
RASH (Skin and subcutaneous tissue disorders) | 20 (23) | 7 (9)
HYPERTENSION (Vascular disorders) | 19 (24) | 27 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No public presentation/publication of any interim results will be made by any principal investigator (PI) or any other member of the study staff without the Sponsor's prior written consent. The PI further agrees to provide to the sponsor 30 days prior to submission, review copies that report any results of the study. The sponsor shall have the right to review, comment, and edit. If the parties disagree, the PI agrees to meet with the sponsor to discuss and resolve any such issues/disagreement.